CLINICAL TRIAL: NCT02015806
Title: Assessing the Impact of Low-Touch Devices on Medication Adherence
Brief Title: Robust Evaluation to Measure Improvements in Nonadherence From Low-cost Devices
Acronym: REMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CVS Caremark (Industry)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-P-00009085
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease; Diabetes; Breast Cancer; Depression; Mental Health Disorder; Prostatic Hypertrophy, Benign; Parkinson's Disease; Epilepsy
Keywords: Quality improvement; Randomized controlled trial; Medication adherence; RxTimer Cap; PillMinder; Take-N-Slide; Low-touch devices; Medication management
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Breast Neoplasms; Depression; Mental Disorders; Prostatic Hyperplasia; Parkinson Disease; Epilepsy; Medication Adherence

ARMS (14):
- All meds but depression, 1x daily use, RxTimerCap (Experimental): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to receive a RxTimerCap.
  Interventions: Behavioral: RxTimerCap
- All meds but depression, 1x daily use, Take-N-Slide (Experimental): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to receive a Take-N-Slide.
  Interventions: Behavioral: Take-N-Slide
- All meds but depression, 1x daily use, pillbox (Experimental): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to receive a standard pillbox.
  Interventions: Behavioral: Pillbox
- All meds but depression, 1x daily use, control (No Intervention): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to continue with usual care.
- All meds but depression, ≥1 med >1 daily use, RxTimerCap (Experimental): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, who have at least one medication that is intended for use more than once daily, and who are randomized to receive a RxTimerCap.
  Interventions: Behavioral: RxTimerCap
- All meds but depression, ≥1 med >1 daily use, pillbox (Experimental): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, who have at least one medication that is intended for use more than once daily, and who are randomized to receive a standard pillbox.
  Interventions: Behavioral: Pillbox
- All meds but depression, ≥1 med >1 daily use, control (No Intervention): Individuals who are taking 1-3 cardiovascular or other non-depression chronic disease medications and who are suboptimally adherent to these therapies, who have at least one medication that is intended for use more than once daily, and who are randomized to continue with usual care.
- Only depression meds, 1x daily use, RxTimerCap (Experimental): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to receive a RxTimerCap.
  Interventions: Behavioral: RxTimerCap
- Only depression meds, 1x daily use, Take-N-Slide (Experimental): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to receive a Take-N-Slide.
  Interventions: Behavioral: Take-N-Slide
- Only depression meds, 1x daily use, pillbox (Experimental): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to receive a standard pillbox.
  Interventions: Behavioral: Pillbox
- Only depression meds, 1x daily use, control (No Intervention): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, whose medications are all intended for once daily use, and who are randomized to continue with usual care.
- Only depression meds, ≥1 med >1 daily use, RxTimerCap (Experimental): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, who have at least one medication that is intended for use more than once daily, and who are randomized to receive a RxTimerCap.
  Interventions: Behavioral: RxTimerCap
- Only depression meds, ≥1 med >1 daily use, pillbox (Experimental): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, who have at least one medication that is intended for use more than once daily, and who are randomized to receive a standard pillbox.
  Interventions: Behavioral: Pillbox
- Only depression meds, ≥1 med >1 daily use, control (No Intervention): Individuals who are taking only antidepressants and who are suboptimally adherent to these therapies, who have at least one medication that is intended for use more than once daily, and who are randomized to continue with usual care.

INTERVENTIONS:
Behavioral: RxTimerCap — The RxTimerCap is a pill bottle cap with a digital timer that shows the time elapsed since the medication was last taken. Patients randomized to receive the RxTimerCap will receive a one-time mailing with one device for each of the maintenance medications they were using at the time of identification for study eligibility; additionally, patients will receive an information card explaining the device's use which includes a telephone number at which they can get additional information.
  Arms: All meds but depression, 1x daily use, RxTimerCap; All meds but depression, ≥1 med >1 daily use, RxTimerCap; Only depression meds, 1x daily use, RxTimerCap; Only depression meds, ≥1 med >1 daily use, RxTimerCap
Behavioral: Take-N-Slide — The Take-N-Slide device is a patented strip with toggles for each day of the week which are meant to be slid after taking a medication. Each Take-N-Slide can be removed and reused for the next prescription bottle. Patients randomized to receive Take-N-Slide will receive a one-time mailing with one device for each of the maintenance medications they were using at the time of identification for study eligibility; additionally, patients will receive an information card explaining the device's use which includes a telephone number at which they can get additional information.
  Arms: All meds but depression, 1x daily use, Take-N-Slide; Only depression meds, 1x daily use, Take-N-Slide
Behavioral: Pillbox — The standard pillbox is a plastic organization box with one compartment for every day of the week. Patients randomized to receive a pillbox will receive a one-time mailing with one device for each of the maintenance medications they were using at the time of identification for study eligibility; additionally, patients will receive an information card explaining the device's use which includes a telephone number at which they can get additional information.
  Arms: All meds but depression, 1x daily use, pillbox; All meds but depression, ≥1 med >1 daily use, pillbox; Only depression meds, 1x daily use, pillbox; Only depression meds, ≥1 med >1 daily use, pillbox

SUMMARY:
The aim of this study is to determine whether adherence to oral maintenance medications differs for patients randomized to receive a RxTimerCap, a Take-N-Slide, a standard pillbox, or none of these devices, with the hypothesis that low-touch devices improve adherence over control and that the increase in adherence is agnostic across devices.

DETAILED DESCRIPTION:
Prior to randomization, all patients meeting the inclusion criteria stratified into two strata and two blocks within each strata. The first stratum will consist of all patients on 1 to 3 medications for cardiovascular or other non-depression chronic conditions who are suboptimally adherent to these therapies. The second stratum will include all patients whose only targeted medications are for depression and who are suboptimally adherent to this therapy. Given that the Take-N-Slide device only has a Yes/No toggle for each day of the week and can therefore only be used once per day, each stratum will be further stratified into two separate blocks based on the frequency with which the study participants' medications are (or could possibly be) taken. Patients who are on a medication that is used more than once daily will be randomized in a 2:1 ratio to receive the RxTimerCap, pillbox, or to continue with usual care. Patients for whom all medications are dosed once daily will be randomized in a 2:1 ratio to receive the Take-N-Slide, RxTimerCap, pillbox, or to continue with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Have 1 to 3 oral maintenance medications for chronic disease in the 12-month period prior to study eligibility evaluation

  * Cardiovascular disease (defined as hypertension, hyperlipidemia, coronary artery disease, congestive heart failure, or diabetes); OR
  * Another non-depression chronic condition (defined as breast cancer, benign prostatic hypertrophy, schizophrenia, bipolar disorder, anxiety, arrythmia; Parkinson's disease, seizure, and epilepsy); OR
  * Depression
* Be suboptimally adherent to their qualifying medications, defined as a Medication Possession Ratio between 30% and 80% during the 12 months preceding identification of study eligibility
* Eligible for pharmacy benefits during the 12 months prior to being identified as being eligible for the study and expected to be eligible for pharmacy benefits through the end of the evaluation period.

Exclusion Criteria:

* Enrolled in Ready Fill at Mail (a pharmacy benefit program whereby members elect to have medications shipped automatically to them at the time of refill due date or prescription renewal).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53480 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Optimal medication adherence to all cardiovascular or non-depression chronic disease medications | 12 months
  Optimal adherence to all cardiovascular or non-depression chronic disease medications, defined as a Medication Possession Ratio (MPR) equal to or greater than 80% and assessed using administrative pharmacy claims

SECONDARY OUTCOMES:
Optimal adherence to antidepressants | 12 months
  Optimal adherence to antidepressants among subjects whose only targeted therapy is an antidepressant, calculated using Medication Possession Ratios (MPR) and assessed using administrative pharmacy claims
Optimal adherence to the targeted therapies in each randomization block independently | 12 months
  Optimal adherence to the targeted therapies in each of the randomization blocks independently, calculated using Medication Possession Ratios (MPR) and assessed using administrative pharmacy claims
Optimal adherence to cardiovascular medications among subjects who are suboptimally adherent to these medications at time of randomization | 12 months
  Optimal adherence to cardiovascular medications among subjects who are suboptimally adherent to these medications at time of randomization, calculated using Medication Possession Ratios (MPR) and assessed using administrative pharmacy claims

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- CVS Health, Woonsocket, Rhode Island, United States

REFERENCES:
- [Derived] Al-Aqeel S, Gershuni O, Al-Sabhan J, Hiligsmann M. Strategies for improving adherence to antiepileptic drug treatment in people with epilepsy. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD008312. doi: 10.1002/14651858.CD008312.pub4. PMID 33089492
- [Derived] Choudhry NK, Krumme AA, Ercole PM, Girdish C, Tong AY, Khan NF, Brennan TA, Matlin OS, Shrank WH, Franklin JM. Effect of Reminder Devices on Medication Adherence: The REMIND Randomized Clinical Trial. JAMA Intern Med. 2017 May 1;177(5):624-631. doi: 10.1001/jamainternmed.2016.9627. PMID 28241271